CLINICAL TRIAL: NCT00695617
Title: Citrate Anticoagulation During MARS Treatment
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Pieter Evenepoel, University Hospitals Leuven
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ML4960
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2009-03-05 (Estimated); Status verified 2009-03

CONDITIONS: Liver Failure
Keywords: MARS treatment; Citrate anticoagulation
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): citrate first
  Interventions: Drug: trisodiumcitrate
- B (Experimental): no anticoagulation first
  Interventions: Drug: trisodiumcitrate

INTERVENTIONS:
Drug: trisodiumcitrate — trisodiumcitrate 1.035 M
  Arms: A
Drug: trisodiumcitrate — trisodiumcitrate 1.035 M
  Arms: B

SUMMARY:
The optimal anticoagulation procedure during MARS treatment has not been defined. In various multi-centre trials, such as MARS-RELIEF, anticoagulation procedures are left to the discretion of the treating physician. On the one hand, given the increased risk of bleeding associated with liver failure, high dosage of anticoagulation therapy should be avoided. On the other hand, contact of blood or blood components with the extracorporeal circuit will likely result in coagulation activation or even loss of coagulation factors.

Citrate anticoagulation has gained popularity, especially in hemodialysis patients. It results in a highly effective anticoagulation, exclusively confined to the extracorporeal circulation. Moreover, dependent on the type of dialyser membrane, citrate anticoagulation resulted in reduced activation of other cellular components.

In contrast to hemodialysis patients, experience with citrate anticoagulation during treatment with artificial liver devices is limited. The liver contributes substantially to the metabolism of exogenous citrate. As a result, cirrhotic patients have decreased endogenous citrate clearances. Importantly, blood purification devices contribute substantially to overall citrate clearance, thereby preventing accumulation of citrate. Several centres, including our own, have gained experience with citrate anticoagulation during fractionated plasma separation and adsorption (FPSA), a related liver dialysis device, in the treatment of liver failure patients.

Citrate anticoagulation during MARS treatment has not been studied so far.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled MARS treatment
* Age over 18 years
* Informed consent
* Admitted to Intensive Care Unit

Exclusion Criteria:

* Blood or plasma transfusion within 48 hours before study
* Hypocalcemia (ionised Ca < 0.90 mmol/l)
* Acidosis (pH < 7.25) due to any cause
* Use of citrate containing medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Extracorporeal circuit coagulation events | 6 hours

SECONDARY OUTCOMES:
Citrate tolerability | 6 hours
Treatment efficacy | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Evenepoel, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Bjorn Meijers, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Alexander Wilmer, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Frederik Nevens, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Meijers BK, Verhamme P, Nevens F, Hoylaerts MF, Bammens B, Wilmer A, Arnout J, Vanrenterghem Y, Evenepoel P. Major coagulation disturbances during fractionated plasma separation and adsorption. Am J Transplant. 2007 Sep;7(9):2195-9. doi: 10.1111/j.1600-6143.2007.01909.x. Epub 2007 Jul 19. PMID 17640311